CLINICAL TRIAL: NCT03207074
Title: Pilot Study: Can the iKnife (Rapid Evaporative Ionisation Mass Spectrometry) Distinguish Between Normal and Malignant Endometrial Tissue?
Brief Title: Can the iKnife Distinguish Between Normal and Malignant Endometrial Tissue?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16HH3687 iKnife EC
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Results first posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-06

CONDITIONS: Endometrial Neoplasms; Endometrial Cancer; Endometrial Hyperplasia; Endometrial Diseases
Keywords: iKnife; Mass Spectrometry; Point-of-care; Diagnosis; Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Hyperplasia; Uterine Diseases; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Other): Single study arm. All patients who participate in the study will receive conventional histological diagnosis and diagnosis with the new technology (iKnife)
  Interventions: Diagnostic Test: iKnife i.e. Rapid Evaporative Ionisation Mass Spectrometry

INTERVENTIONS:
Diagnostic Test: iKnife i.e. Rapid Evaporative Ionisation Mass Spectrometry — The endometrial tissue will be analysed by this new technology and compared to gold standard (histopathology)

SUMMARY:
Aim: Determine if Rapid Evaporative Ionization Mass Spectrometry (the iKnife); can diagnose cancer and pre-cancer from endometrial tissue biopsy samples.

Women attending a gynaecology clinic for assessment of abnormal bleeding will receive an pelvic (internal) ultrasound as routine standard of care. If any abnormalities are detected, a tissue sample will be needed. If women are agreeable a second tissue sample will be taken for research. The first will be analysed by conventional means (histopathology). The second sample with new technology called the 'iKnife'. This is a modified type of Mass spectrometry device, that separates particles based on their mass charge ratio. The idea being that if tissue is burnt, gas is produced, and this gas contains lots of ions that can be analysed by the iKnife. Each type of tissue (cancer or non-cancer) will have a unique signature that the iKnife can use to distinguish between samples. If effective it could be used in future outpatient clinics to provide a one-stop, true point of care diagnosis.

DETAILED DESCRIPTION:
Aim: Determine if Rapid Evaporative Ionization Mass Spectrometry (the iKnife); can diagnose cancer and pre-cancer from endometrial tissue biopsy samples.

Background:

Endometrial cancer is a tumour originating in the endometrium (womb lining); it is the most common gynaecological cancer in the United Kingdom (UK). In 2012, there were almost 100,000 new cases diagnosed in Europe. Endometrial cancer classically presents with postmenopausal bleeding (bleeding after the menopause), or intermenstrual bleeding (bleeding between periods).

Although routine management for these women does vary, in general a screening test is performed, typically a pelvic (internal) ultrasound to assess the endometrium (womb lining). In cases where the endometrial thickness is above the threshold for investigation -an endometrial biopsy (sampling cells from the womb lining) is indicated.

Once the endometrial biopsy is performed, it is sent to the histologist for further examination. Histological analysis may take several days and patients are either brought back to clinic for discussion of the results or are given a telephone appointment. The patient often will not know the result of the test for up to 2 weeks; thus causing a lot of unnecessary anxiety and distress. Novel diagnostic tests, such as Rapid Evaporative Ionization Mass Spectrometry (REIMS), may enable real time point of care diagnosis for the first time. When REIMS is coupled to conventional surgical diathermy it is colloquially referred to as the iKnife. REIMS has been used successfully in other organs and has been shown to accurately distinguish between cancer and non-cancer. Part of this research project is to evaluate this new technology in endometrial cancer.

The study:

All women presenting to the rapid access clinic with post menopausal bleeding (PMB) and intermenstrual bleeding will be approached for consent for inclusion into this study. They will receive the patient information leaflet when they arrive in clinic and are waiting to see the clinician. When women normally attend this clinic the doctor will discuss what will happen - this includes an internal (pelvic scan) and an examination. If the womb lining is thickened on the scan the patient will need a tissue biopsy (this is not that common, most women only need a scan), this will be taken at the same time as the examination in clinic. The device used to take the tissue biopsy is called a pipelle. It is a fine 3mm width tube with suction which removes cells from the lining of the womb. If the patient is agreeable a second endometrial sample will be taken specifically for research.

The histology of first sample will be analysed by conventional pathology and the second sample will be analysed by the new technology REIMS. REIMS is Rapid Evaporative Ionization Mass Spectrometry. This new technology uses mass spectroscopy to analyse the tissue. REIMS has been dubbed the 'iKnife' or 'intelligent knife' colloquially as when coupled with surgical diathermy the gas pattern produced is unique to the tissue and helps surgeons know where to cut. The diagnostic ability of this technology will be compared against the gold standard, which is histological examination.

Patients who already have a diagnosis of endometrial cancer and can still participate in the study if they are undergoing a hysterectomy, as can consent to an tissue biopsy sample in theatre (either under general anaesthesia, GA or ex-vivo).

If this technology proves effective it will mean that womb (endometrial) cancer can be diagnosed from samples taken in clinic on the same day; providing a true one stop clinic, for the first time.

ELIGIBILITY:
Inclusion Criteria:

* All women presenting to rapid access gynaecology clinic with postmenopausal bleeding or intermenstrual bleeding or referred with a confirmed diagnosis of endometrial cancer.

Exclusion Criteria:

* Anyone lacking capacity. <18years old. Pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study is looking at endometrial cancer so recruitment of women only
Enrollment: 150 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Charlotte and Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients attending rapid access clinic, or day surgery for investigation of suspected endometrial cancer were asked to participate in the study. Those needing tissue biopsies for clinical indications, were also asked to undergo a second research biopsy. The research biopsy is analysed by the iKnife.
Groups:
- All Patients: Single study arm. All patients who participate in the study will receive a tissue biopsy, one processed with the conventional histology and one processed with the iKnife (Rapid Evaporative Ionisation Mass Spectrometry).
Period: Overall Study
Arm/Group | All Patients
Started | 150
Completed | 150
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 150
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.7 (8.4)

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Ability of iKnife (REIMS) in Detection of Cancer and Pre-cancer in Endometrial Biopsy Specimens
Description: Sensitivity, specificity and positive and negative predictive values will be obtained for this new technology compared to gold standard (histopathological exam).
  Test sensitivity is the ability of the iknife to correctly identify those with endometrial cancer (true positive rate).
  Test specificity is the ability of the iKnife to correctly identify those without endometrial cancer (true negative rate).
  Positive predictive value is the probability that patients with a positive iKnife test result truly have the disease.
  Negative predictive value is the probability that patients with a negative screening iKnife test truly don't have endometrial cancer.
Time Frame: Each patient was assessed in clinic and the research biopsy was performed during the clinic visit. It was processed within 4 hours by the iKnife (or snap frozen and processed at a later date, within 3months)
Population: Analysis of diagnostic accuracy of iKnife from endometrial pipelle biopsies
Measure: Number; unit: percentage
Arm/Group | All Patients
Number analyzed (Participants) | 150
percentage
  Sensitivity | 79
  Specificity | 96
  Positive Predictive value | 93
  Negative predictive value | 86

ADVERSE EVENTS:
Time Frame: The duration of study collection June 2017-June 2019, (2 years). Adverse events such as perforation, if they were to occur would happen only at the time of biopsy therefore the risk was within 24 hours of the biopsy.
Description: The patients provided a tissue biopsy sample for research (in addition to the tissue sample provided for clinical indications).
  No extra additional risk for the patient. However, tissue biopsy can be inadequate, or can cause perforation (1-2%). There is negligable additional risk with the extra research tissue needed.
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 0/150
Serious Adverse Events (participants affected / at risk) | 0/150
Other Adverse Events (participants affected / at risk) | 0/150

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT03207074/Prot_SAP_000.pdf